CLINICAL TRIAL: NCT01325909
Title: Does Short-term Exercise Intervention Improve Pre-operative Physical Fitness Following Neoadjuvant Chemoradiotherapy in Colorectal Cancer Patients?
Brief Title: Exercise Training in Colorectal Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michelle Mossa (Other Government)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, Michelle Mossa, Research and Development Director, Liverpool University Hospitals NHS Foundation Trust
Organization: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 11/H1002/12
Record Dates: First submitted 2011-03-29; First posted 2011-03-30 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Active Comparator)
  Interventions: Behavioral: Exercise programme
- No Exercise (No Intervention)

INTERVENTIONS:
Behavioral: Exercise programme
  Arms: Exercise

SUMMARY:
Neoadjuvant chemoradiotherapy (NACRT) prior to surgery for lower gastrointestinal (colon and rectal) cancer is associated with improved survival, but also adversely affects physical fitness, potentially rendering patients unfit for major surgery or increasing the risk of adverse outcome (death and serious complications) after major surgery. The investigators have pilot data using an upper gastrointestinal cancer patient cohort showing that neoadjuvant chemotherapy (NAC)reduces objectively measured exercise capacity (fitness). The investigators therefore propose a blinded, single centre, prospective interventional trial of patients undergoing NACRT prior to elective colorectal cancer resection in an NHS teaching hospital.

The investigators wish to explore various hypotheses:

1. Is exercise intervention feasible and tolerable in this cohort of patients?
2. Can fitness be improved using a structured, responsive exercise training programme (SRETP)?
3. Can SRETP improve quality of life?
4. Can SRETP improve physical activity?
5. Can SRETP improve surgical outcome?
6. Can physiological fitness and oncological outcome be matched to identify an optimal time for physiological recovery following NACRT prior to major surgery.

The investigators aim to recruit 5 patients for a feasibility and tolerably study and 30 patients for an interventional study over 24 months from Aintree University Teaching Hospitals NHS Foundation Trust. Consenting patients will undergo a series of tests designed to evaluate the ability of the muscle to take up and utilise oxygen, namely a cardiopulmonary exercise test (CPET) and VO2 Kinetics tests, all done pre-CRT and at 3,6,9 and 14 weeks post-CRT (pre-surgery). All patients will have their CPET, as well as standard restaging scans at 9 and 14 weeks post NACRT. Outcome, activity and quality of life data will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* All patients listed to undergo elective colorectal cancer resection and longcourse neoadjuvant chemoradiotherapy at Aintree University Hospitals NHS Foundation Trust

Exclusion Criteria:

* Unable to consent
* Under 18 years of age
* Unable to perform exercise
* Meet any contraindications on the ATS CPET safety guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Maintain or improve physical fitness (anaerobic threshold measured by CPET)after treatment with neoadjuvant chemoradiotherapy in colorectal cancer patients. | 3 years

SECONDARY OUTCOMES:
Other measures of physical fitness measured in CPET or the VO2 kinetics test | 3 years
Adherence to a 6 week interval exercise intervention. | 3 years
Optimal time for surgery indicating optimal oncological and physiological fitness | 3 years
Health related quality of life improvement as measured by SF36, EORCT c30 v3 | 3 years
Outcome from major surgery measured by 5 day POMS | 3 years
Activity levels before during and after neoadjuvant chemoradiotherapy | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm A West, MD MRCS, Principal Investigator — Aintree University Hospitals NHS Foundation Trust, Liverpool, UK
Locations (1):
- Aintree University Hospitals, Liverpool, United Kingdom

REFERENCES:
- [Derived] Loughney L, West MA, Dimitrov BD, Kemp GJ, Grocott MP, Jack S. Physical activity levels in locally advanced rectal cancer patients following neoadjuvant chemoradiotherapy and an exercise training programme before surgery: a pilot study. Perioper Med (Lond). 2017 Feb 16;6:3. doi: 10.1186/s13741-017-0058-3. eCollection 2017. PMID 28228938
- [Derived] Brunet J, Burke S, Grocott MP, West MA, Jack S. The effects of exercise on pain, fatigue, insomnia, and health perceptions in patients with operable advanced stage rectal cancer prior to surgery: a pilot trial. BMC Cancer. 2017 Feb 23;17(1):153. doi: 10.1186/s12885-017-3130-y. PMID 28228123
- [Derived] West MA, Dimitrov BD, Moyses HE, Kemp GJ, Loughney L, White D, Grocott MP, Jack S, Brown G. Timing of surgery following neoadjuvant chemoradiotherapy in locally advanced rectal cancer - A comparison of magnetic resonance imaging at two time points and histopathological responses. Eur J Surg Oncol. 2016 Sep;42(9):1350-8. doi: 10.1016/j.ejso.2016.04.003. Epub 2016 Apr 26. PMID 27160356
- [Derived] West MA, Loughney L, Lythgoe D, Barben CP, Sripadam R, Kemp GJ, Grocott MP, Jack S. Effect of prehabilitation on objectively measured physical fitness after neoadjuvant treatment in preoperative rectal cancer patients: a blinded interventional pilot study. Br J Anaesth. 2015 Feb;114(2):244-51. doi: 10.1093/bja/aeu318. Epub 2014 Oct 1. PMID 25274049